CLINICAL TRIAL: NCT00618813
Title: A Pilot Study of Chemotherapy Intensification by Adding Vincristine, Topotecan and Cyclophosphamide to Standard Chemotherapy Agents With an Interval Compression Schedule in Newly Diagnosed Patients With Localized Ewing Sarcoma Family of Tumors
Brief Title: Two Regimens of Combination Chemotherapy in Treating Younger Patients With Newly Diagnosed Localized Ewing Sarcoma Family of Tumors
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Children's Oncology Group (Network)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: AEWS07P1; NCI-2009-00371 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); CDR0000586282 (Other: Clinical Trials.gov); U10CA098543 (NIH); COG-AEWS07P1 (Other: Children's Oncology Group)
Record Dates: First submitted 2008-02-19; First posted 2008-02-20 (Estimated); Results first posted 2014-02-10 (Estimated); Last update posted 2014-09-25 (Estimated); Status verified 2014-09

CONDITIONS: Ewing Sarcoma of Bone; Localized Ewing Sarcoma/Peripheral Primitive Neuroectodermal Tumor
MeSH Terms: conditions — Neuroectodermal Tumors, Primitive, Peripheral | interventions — Radiotherapy; Radiation; Etoposide; Ifosfamide; indolepropanol phosphate; Doxorubicin; Cyclophosphamide; Vincristine; Topotecan; trioctyl phosphine oxide; Filgrastim; Granulocyte Colony-Stimulating Factor

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Treatment (combination chemotherapy) (Experimental): See Detailed Description
  Interventions: Other: radiation therapy; Other: therapeutic conventional surgery; Drug: etoposide; Drug: ifosfamide; Drug: doxorubicin hydrochloride; Drug: cyclophosphamide; Drug: vincristine sulfate; Drug: topotecan hydrochloride; Biological: filgrastim

INTERVENTIONS:
Other: radiation therapy — Undergo radiation therapy
  Other Names: irradiation; radiotherapy; therapy, radiation
Other: therapeutic conventional surgery — Undergo surgery
Drug: etoposide — Given IV
  Other Names: EPEG; VP-16; VP-16-213
Drug: ifosfamide — Given IV
  Other Names: Cyfos; Holoxan; IFF; IFX; IPP
Drug: doxorubicin hydrochloride — Given IV
  Other Names: ADM; ADR; Adria; Adriamycin PFS; Adriamycin RDF
Drug: cyclophosphamide — Given IV
  Other Names: CPM; CTX; Cytoxan; Endoxan; Endoxana
Drug: vincristine sulfate — Given IV
  Other Names: leurocristine sulfate; VCR; Vincasar PFS
Drug: topotecan hydrochloride — Given IV
  Other Names: hycamptamine; Hycamtin; SKF S-104864-A; TOPO
Biological: filgrastim — Given SC
  Other Names: G-CSF; Neupogen

SUMMARY:
This clinical trial is studying the side effects of combination chemotherapy and to see how well they work in treating patients with newly diagnosed localized Ewing sarcoma family of tumors. Drugs used in chemotherapy work in different ways to stop the growth of tumor cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) and giving the drugs in different ways may kill more tumor cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To assess the feasibility and safety of adding interval-compressed vincristine, topotecan hydrochloride, and cyclophosphamide to a treatment protocol utilizing interval compression of vincristine, doxorubicin hydrochloride, cyclophosphamide, ifosfamide, and etoposide in patients with localized Ewing sarcoma family of tumors.

SECONDARY OBJECTIVES:

I. To estimate the event-free survival in patients treated with this regimen.

OUTLINE: This is a multicenter study.

INDUCTION THERAPY (WEEKS 1-12): Patients receive vincristine IV on day 1 in weeks 1, 2, 5, 6, 9, 10, 11, and 12; topotecan hydrochloride IV over 30 minutes on days 1-5 in weeks 1 and 9; cyclophosphamide IV over 1 hour on days 1-5 in weeks 1 and 9 and on day 1 in weeks 5 and 11; ifosfamide IV over 1 hour on days 1-5 in weeks 3 and 7; etoposide IV over 1 hour on days 1-5 in weeks 3 and 7; and doxorubicin hydrochloride IV over 15 minutes on days 1 and 2 in weeks 5 and 11. Patients also receive filgrastim (G-CSF) subcutaneously (SC) beginning 24-36 hours after the last dose of chemotherapy and continuing for at least 7 days or until blood counts recover, whichever comes last. Filgrastim is discontinued at least 24 hours prior to the next course of chemotherapy.

LOCAL CONTROL: Patients who respond to induction therapy may undergo surgery alone if the lesion can be resected with negative margins and with a reasonable functional result beginning in week 13. Following surgery, patients with unresectable lesions or inadequate margins may receive radiotherapy during week 15. Patients with bulky lesions in surgically difficult sites such as the spine, skull, and periacetabular pelvis; poor response to induction chemotherapy; or those in whom surgery would result in unacceptable functional results may receive radiotherapy alone in weeks 13-19. Patients with bulky lesions in difficult sites and who do not have a good clinical and radiographic response to induction therapy may receive radiotherapy to the primary site during weeks 13-19 followed by surgery of the involved site during week 25 after recovery from course 11 of chemotherapy. Patients with microscopic residual disease after planned pre-operative radiotherapy will receive additional radiotherapy.

CONTINUATION THERAPY (WEEKS 15-36): Patients receive vincristine IV on day 1 in weeks 15, 16, 21-24, 27-30, 33, and 34; topotecan hydrochloride IV over 30 minutes on days 1-5 in weeks 15, 21, and 29; cyclophosphamide IV over 1 hour on days 1-5 in weeks 15, 21 and 29 and on day 1 in weeks 23, 27, and 33; ifosfamide IV over 1 hour on days 1-5 in weeks 17, 19, 25, 31, and 35; etoposide IV over 1 hour on days 1-5 in weeks 17, 19, 25, 31, and 35; and doxorubicin hydrochloride IV over 15 minutes on days 1 and 2 of weeks 23, 27, and 33. Patients also receive G-CSF SC as in induction therapy.

After completion of study treatment, patients are followed for 10 years.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of extracranial Ewing sarcoma or peripheral primitive neuroectodermal tumor of bone or soft tissue:

  * Newly diagnosed disease
  * Disease confirmed by biopsy only with no attempt at complete or partial resection

    * Unplanned excision allowed provided adequate imaging was obtained prior to surgery and incompletely resected disease is controlled by local therapy
  * No esthesioneuroblastoma
* Localized disease, including any of the following sites:

  * Chest wall tumors with ipsilateral pleural effusions, ipsilateral positive pleural fluid cytology, or ipsilateral pleural based secondary tumor nodules;

    * No contralateral pleural effusions or pleural nodules
  * Regional lymph nodes that are clinically suspicious or confirmed by biopsy

    * No distant lymph node metastases
  * Extra-dural tumors arising in the bony skull

    * No tumors arising in the intra-dural soft tissue or the intra-dural region of the spine
* No evidence of metastatic disease, defined as any of the following:

  * Lesions that are discontinuous from the primary tumor
  * Lesions that are not regional lymph nodes
  * Lesions that do not share a body cavity with the primary tumor
* No evidence by CT scan of metastatic lung disease, defined as any of the following:

  * One pulmonary nodule > 1 cm in diameter or more than one nodule > 0.5 cm diameter

    * Pulmonary nodules that are resected and are not found to be metastatic Ewing sarcoma are allowed
  * Biopsy proven solitary nodules measuring 0.5 to 1.0 cm or multiple nodules measuring 0.3 to 0.5 cm

    * Solitary nodules measuring < 0.5 cm or multiple nodules measuring < 0.3 cm are allowed unless biopsy proven to be metastatic (biopsy is not required)
* Karnofsky performance status (PS) 0-2 (>= 16 years old) OR Lansky PS 0-2 (< 16 years old)
* Creatinine clearance or radioisotope glomerular filtration rate ≥ 70 mL/min OR serum creatinine based on age/gender as follows:

  * 1 month to < 6 months old (males and females 0.4 mg/dL)
  * 6 months to < 1 year old (males and females 0.5 mg/dL)
  * 1 to < 2 years old (males and females 0.6 mg/dL)
  * 2 to < 6 years old (males and females 0.8 mg/dL)
  * 6 to < 10 years old (males and females 1.0 mg/dL)
  * 10 to < 13 years old (males and females 1.2 mg/dL)
  * 13 to < 16 years old (males 1.5 mg/dL and females 1.4 mg/dL)
  * >= 16 years old (males 1.7 mg/dL and females 1.4 mg/dL)
* AST or ALT < 2.5 times ULN for age
* Total bilirubin =< 1.5 times upper limit of normal (ULN) for age
* Shortening fraction of >= 27% by ECHO or ejection fraction of >= 50% by radionuclide angiogram (MUGA)
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception
* No prior chemotherapy or radiotherapy
* No concurrent pegfilgrastim (Neulasta) or sargramostim (GM-CSF)
* No other concurrent cancer chemotherapy or immunomodulating agents, including steroids, unless used as an antiemetic

Max Age: 30 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 35 (Actual)
Dates: Start 2008-03; Primary Completion 2010-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Leo Mascarenhas, MD MS, Principal Investigator — Children's Oncology Group
Locations (1):
- Children's Oncology Group, Monrovia, California, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Treatment (Combination Chemotherapy)
Started | 35
Completed Enrollment - Week 12 Treatment | 35 (Patients that complete this segment of protocol therapy are evaluated for outcome measure.)
Completed Week 13 to Week 22 Treatment | 34 (Patients that complete this segment of protocol therapy are evaluated for outcome measure.)
Completed Week 23 to Week 28 Therapy | 34 (Patients that complete this segment of protocol therapy are evaluated for outcome measure.)
Completed Week 29 to Week 37 Therapy | 33 (Patients that complete this segment of protocol therapy are evaluated for outcome measure.)
Completed | 31
Not Completed | 4
Not completed — Lack of Efficacy | 1
Not completed — Physician Decision | 2
Not completed — Withdrawal by Subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 35
Age, Continuous [Median (Full Range); unit: years] | 11 [0 to 22]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 16
  Male | 19
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 10
  Not Hispanic or Latino | 25
  Unknown or Not Reported | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 0
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 29
  More than one race | 0
  Unknown or Not Reported | 6
Region of Enrollment [Number; unit: participants]
  United States | 33
  Canada | 1
  Australia | 1

OUTCOME MEASURES:

1. Primary Outcome: Incidence of Death
Description: Incidence of death from complications of therapy while the patient is on protocol therapy or within one month of terminating protocol therapy
Time Frame: Length of protocol therapy (up to 37 weeks) plus 30 days
Population: Any patient who receives at least one cycle of protocol therapy, or who dies as a result of complications of therapy prior to completing one cycle of therapy will be evaluable for this outcome
Measure: Number; unit: participants
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 35
participants | 0

2. Primary Outcome: Incidence Rate (Number of Participants) of Dose-limiting Toxicity (DLT) - Enrollment to Week 12
Description: The incidence rate of DLT while on protocol therapy where DLT is defined as (1) Grade 3 or greater nonhematological adverse event that is possibly, probably, or likely related to therapy with the specific exception of Grade 3 or greater nausea or vomiting controlled by standard supportive care measures, Grade 3 infection and Grade 3 alopecia; or (2) Grade 4 or higher hematological AE that delays the administration of therapy at least 2 weeks.
Time Frame: Enrollment to week 12
Population: Any patient who receives at least one cycle of protocol therapy, or who is removed from protocol therapy partly or solely because of a dose-limiting toxicity will be evaluable for this outcome.
Measure: Number; unit: participants
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 35
participants | 12

3. Primary Outcome: Incidence Rate (Number of Participants) of Dose-limiting Toxicity (DLT) - Week 13 to Week 22
Description: as for outcome 2
Time Frame: Week 13 to week 22
Population: One patient was not evaluated for dose-limiting toxicity during weeks 13-22 because patient did not complete that segment of protocol therapy.
Measure: Number; unit: participants
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 34
participants | 9

4. Primary Outcome: Incidence Rate (Number of Participants) of Dose-limiting Toxicity (DLT) - Week 23 to Week 28
Description: as for outcome 2
Time Frame: Week 23 to week 28
Population: One patient was not evaluated for DLT during weeks 23-28 because the patient did not complete that segment of therapy.
Measure: Number; unit: participants
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 34
participants | 9

5. Primary Outcome: Incidence Rate (Number of Participants) of Dose-limiting Toxicity (DLT) - Week 29 to Week 37
Description: as for outcome 2
Time Frame: Week 29 to week 37
Population: Two patients were not evaluated for DLT during weeks 29-37 because those patients did not complete that segment of protocol therapy.
Measure: Number; unit: participants
Arm/Group | Treatment (Combination Chemotherapy)
Number analyzed (Participants) | 33
participants | 14

6. Secondary Outcome: Event Free Survival
Description: Disease progression, occurrence of a second malignant neoplasm (SMN)or death will be considered an analytic event. In all other cases, the patient will be considered censored at last contact.
Time Frame: From enrollment to event or 10 years from enrollment, whichever occurs first
Reporting Status: Not Posted

ADVERSE EVENTS:
Description: One patient was not evaluated for DLT during weeks 13-22 and 23-28 because patient did not complete that segment of therapy. Two patients were not evaluated for DLT during weeks 29-37 because they did not complete that segment of therapy.
Arm/Group | Treatment (Combination Chemotherapy)
Serious Adverse Events (participants affected / at risk) | 2/35
Other Adverse Events (participants affected / at risk) | 33/35
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Combination Chemotherapy) (N=35)
Anemia (Blood and lymphatic system disorders) | 1
Apnea (Respiratory, thoracic and mediastinal disorders) | 1
Platelet count decreased (Investigations) | 1
Upper gastrointestinal hemorrhage (Gastrointestinal disorders) | 1
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Treatment (Combination Chemotherapy) (N=35)
Abdominal pain (Gastrointestinal disorders) | 4
Alanine aminotransferase increased (Investigations) | 6
Anemia (Blood and lymphatic system disorders) | 25
Anorectal infection (Infections and infestations) | 1
Anorexia (Metabolism and nutrition disorders) | 3
Anxiety (Psychiatric disorders) | 1
Apnea (Respiratory, thoracic and mediastinal disorders) | 1
Appendicitis (Infections and infestations) | 1
Aspartate aminotransferase increased (Investigations) | 1
Back pain (Musculoskeletal and connective tissue disorders) | 1
Bladder infection (Infections and infestations) | 1
Blood bilirubin increased (Investigations) | 1
Constipation (Gastrointestinal disorders) | 1
Dehydration (Metabolism and nutrition disorders) | 1
Depression (Psychiatric disorders) | 1
Dermatitis radiation (Injury, poisoning and procedural complications) | 2
Diarrhea (Gastrointestinal disorders) | 1
Dysphagia (Gastrointestinal disorders) | 1
Encephalopathy (Nervous system disorders) | 2
Enterocolitis infectious (Infections and infestations) | 2
Esophagitis (Gastrointestinal disorders) | 1
Febrile neutropenia (Blood and lymphatic system disorders) | 17
Fever (General disorders) | 2
Gallbladder obstruction (Hepatobiliary disorders) | 1
Headache (Nervous system disorders) | 2
Hyperglycemia (Metabolism and nutrition disorders) | 4
Hypocalcemia (Metabolism and nutrition disorders) | 2
Hypokalemia (Metabolism and nutrition disorders) | 9
Hypomagnesemia (Metabolism and nutrition disorders) | 1
Hyponatremia (Metabolism and nutrition disorders) | 3
Hypophosphatemia (Metabolism and nutrition disorders) | 4
Hypoxia (Respiratory, thoracic and mediastinal disorders) | 1
Infections and infestations - Other (Infections and infestations) | 18
Intraoperative arterial injury (Injury, poisoning and procedural complications) | 1
Intraoperative neurological injury (Injury, poisoning and procedural complications) | 1
Lung infection (Infections and infestations) | 2
Lymphocyte count decreased (Investigations) | 12
Mucositis oral (Gastrointestinal disorders) | 2
Nausea (Gastrointestinal disorders) | 2
Neutrophil count decreased (Investigations) | 27
Pain (General disorders) | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 1
Perineal pain (Reproductive system and breast disorders) | 1
Peripheral motor neuropathy (Nervous system disorders) | 3
Peripheral sensory neuropathy (Nervous system disorders) | 1
Platelet count decreased (Investigations) | 27
Rectal pain (Gastrointestinal disorders) | 1
Tracheitis (Infections and infestations) | 1
Typhlitis (Gastrointestinal disorders) | 2
Urinary retention (Renal and urinary disorders) | 1
Urinary tract infection (Infections and infestations) | 3
Vomiting (Gastrointestinal disorders) | 1
Weight loss (Investigations) | 1
White blood cell decreased (Investigations) | 26

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Must obtain prior Sponsor approval.